CLINICAL TRIAL: NCT04912596
Title: A Randomized, Single-dose, Double-blind, Double-dummy, Placebo and Active Controlled, Crossover Design Study Using Bronchoprovocation to Evaluate the Pharmacodynamic Equivalence of the Test and Reference Metered Dose Inhalers (MDIs) Containing Albuterol Sulfate in Adult Patients With Stable Mild Asthma
Brief Title: Pharmacodynamic Equivalence of the Test and Reference Metered Dose Inhalers (MDIs) Containing Albuterol Sulfate in Adult Patients With Stable Mild Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: TW20-4643
Record Dates: First submitted 2021-05-28; First posted 2021-06-03 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Mild Asthma
MeSH Terms: interventions — Albuterol; Methacholine Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo group (Placebo Comparator): Two different Reference Placebo inhalers and two different Test Placebo inhalers
  Interventions: Other: Proair HFA or FDA authorized generic: Albuterol Sulfate HFA Inhalation Placebo; Other: Albuterol Sulfate inhalation Placebo; Other: Methacholine
- Reference 1 group (Active Comparator): One Reference inhaler, one Reference Placebo inhaler, and two different Test Placebo inhalers
  Interventions: Drug: Proair HFA (Albuterol Sulfate) or FDA authorized generic: Albuterol Sulfate HFA (Teva Pharmaceutical USA, Inc.) Inhalation Aerosol 108 mcg per actuation; Other: Proair HFA or FDA authorized generic: Albuterol Sulfate HFA Inhalation Placebo; Other: Albuterol Sulfate inhalation Placebo; Other: Methacholine
- Reference 2 group (Active Comparator): Two different Reference inhalers and two different Test Placebo inhalers
  Interventions: Drug: Proair HFA (Albuterol Sulfate) or FDA authorized generic: Albuterol Sulfate HFA (Teva Pharmaceutical USA, Inc.) Inhalation Aerosol 108 mcg per actuation; Other: Albuterol Sulfate inhalation Placebo; Other: Methacholine
- Test group (Experimental): One Test inhaler, one Test Placebo inhaler, and two different Reference Placebo inhalers
  Interventions: Drug: Albuterol Sulfate inhalation aerosol 108 mcg per actuation; Other: Proair HFA or FDA authorized generic: Albuterol Sulfate HFA Inhalation Placebo; Other: Albuterol Sulfate inhalation Placebo; Other: Methacholine

INTERVENTIONS:
Drug: Albuterol Sulfate inhalation aerosol 108 mcg per actuation — equal to albuterol 90 mcg/puff, MDI
  Other Names: Albuterol Sulfate
  Arms: Test group
Drug: Proair HFA (Albuterol Sulfate) or FDA authorized generic: Albuterol Sulfate HFA (Teva Pharmaceutical USA, Inc.) Inhalation Aerosol 108 mcg per actuation — equal to albuterol 90 mcg/puff, MDI
  Other Names: Albuterol Sulfate
  Arms: Reference 1 group; Reference 2 group
Other: Proair HFA or FDA authorized generic: Albuterol Sulfate HFA Inhalation Placebo — MDI
  Arms: Placebo group; Reference 1 group; Test group
Other: Albuterol Sulfate inhalation Placebo — MDI
Other: Methacholine — Methacholine 100 mg/vial

SUMMARY:
The objective of this study is to evaluate the pharmacodynamic (PD) bioequivalence (BE) of albuterol inhalers, test formulation: Albuterol Sulfate HFA inhalation aerosol 108 mcg (equal to albuterol base 90 mcg) per actuation and reference formulation: ProAir HFA (albuterol sulfate) or FDA authorized generic: Albuterol Sulfate HFA (Teva Pharmaceutical USA, Inc.) Inhalation Aerosol 108 mcg (equal to albuterol base 90 mcg) per actuation manufactured by two different manufacturers using methacholine bronchoprovocation challenge test in patients with stable mild asthma.

DETAILED DESCRIPTION:
This study will be conducted using the single-dose, randomized, double-blind, double-dummy, four-sequence, four-treatment, and multiple-center study design to evaluate the PD bioequivalence between the test albuterol sulfate (T) inhalation aerosol 108 mcg per actuation (eq. to albuterol base 90 mcg/puff) and the reference albuterol sulfate (R) (ProAir HFA or FDA authorized generic: Albuterol Sulfate HFA [Teva Pharmaceutical USA, Inc.]) inhalation aerosol 108 mcg per actuation (equal to albuterol base 90 mcg/puff). The two products will be studied using a crossover design in patients with stable mild asthma by administering a minimum of 3 doses of reference product (0, 90, 180 mcg albuterol) and 2 doses of test product (0, 90 mcg albuterol). The bronchodilation potency of albuterol sulfate are measured by the inhibition effects of methacholine challenge on the bronchodilation, as indicated by increase in the provocative concentration of methacholine required to produce a 20% decrease in FEV1 (PC20).

ELIGIBILITY:
Inclusion Criteria:

1. Male, non-pregnant and non-lactating female subjects (20-65 years of age, inclusive).
2. A clinical diagnosis of mild asthma with historical documentation of the asthma diagnosis according to either: (1) the National Asthma Education and Prevention Program (NAEPP) guidelines (2007) or (2) the Global Initiative for Asthma (GINA) Global Strategy for Asthma Management and Prevention (2020).
3. Stable mild asthma receiving the following required inhaled medications for at least 1 month prior to screening: Low doses of ICS alone, or in combination with SABA, used regularly with a stable regimen.
4. Forced Expiratory Volume in 1 second (FEV1) ≥ 80% of the local predicted normal value after withholding SABA ≥ 8 hours.
5. Airway responsiveness to methacholine demonstrated by a pre-albuterol-dose (baseline) PC20 ≤ 8 mg/mL.
6. Nonsmoker for at least 6 months prior to the study and a maximum smoking history of 5 pack-years (the equivalent of one pack per day for 5 years).
7. Provision of written informed consent.
8. Other than asthma, in general good health.
9. Body mass index (BMI) between 17 and 35 kg/m2 (inclusive).
10. Able to correctly use MDI inhalers.
11. Able to perform valid and reproducible pulmonary function tests including no evidence of spirometry effort-induced bronchoconstriction.
12. If the subject or subject's partner is of child-bearing potential, a medically acceptable form of contraception will be used for the duration of the study. Medically acceptable contraceptives include: (1) surgical sterilization, (2) Health Authority approved female hormonal contraceptives, (3) an intrauterine device (IUD), (4) condoms with spermicide, or (5) diaphragm with spermicide.

Exclusion Criteria:

1. Evidence of conditions altering airway reactivity to methacholine, including upper or lower respiratory tract infections (e.g., pneumonia, viral bronchitis, allergic rhinitis, sinobronchitis, etc.) within 6 weeks before Screening.
2. Evidence of a baseline FEV1 < 60% of the local predicted normal value or FEV1 < 1.5 L.
3. History of seasonal asthma exacerbations, in which case the subject should be studied outside of the relevant allergen season.
4. History of cystic fibrosis, bronchiectasis, COPD, or other respiratory diseases including COPD, chronic bronchitis, emphysema, tuberculosis, pulmonary carcinoma, pulmonary fibrosis, pulmonary hypertension that, in the opinion of the Investigator, would compromise subject safety or interfere with the evaluations.
5. History of cardiovascular, hematological, renal, neurologic, hepatic, psychiatric, endocrine dysfunction, including ECG with evidence of ischemic heart diseases and significant arrhythmias.
6. Treatment in an emergency room or hospitalization for acute asthmatic symptoms within 3 months prior to screening.
7. Known intolerance or hypersensitivity to any component of the albuterol MDI, beta2 receptor-agonist drug, HFA, any related compounds or methacholine.
8. Need for daily oral corticosteroids within 3 months prior to screening.
9. Cardiac arrhythmia or 12-lead electrocardiogram (ECG) abnormalities, that in the opinion of the Investigator would compromise subject safety or interfere with the evaluations, or a QTc > 440 ms for males and > 460 ms for females using Fredericia formula.
10. Subjects receiving beta blocker via any route or who may require beta blockers during the study.
11. History of narrow angle glaucoma, convulsive disorders, hyperthyroidism, uncontrolled diabetes, paradoxical bronchospasm.
12. History of malignancies.
13. History of alcohol or drug abuse.
14. Eye, brain, thoracic, and abdominal surgeries within 3 months prior to screening.
15. Use of cromyolyn, leukotriene receptor antagonists (LTRA), nedocromil, zileuton, theophylline, or long-acting beta-agonists (LABA) within 1 month prior to screening.
16. History of receiving muscarinic beta2-agonists (MABAs), short-acting muscarinic antagonists (SAMAs), long-acting muscarinic antagonists (LAMAs), anti-IgE, anti-IL5/5R, anti-IL4R, high dose ICS, or systemic corticosteroid for treatment of asthma within 6 months prior to screening.
17. Known Human Immunodeficiency Virus (HIV)-positive status.
18. Participated in any interventional clinical trials within 1 month prior to screening.
19. Pregnancy or breast feeding.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Post-dose PC20 Concentration | 15 minutes post-dose
  Post-dose PC20, which are the provocative concentrations, respectively, of the methacholine challenge agent required to reduce the forced expiratory volume in one second (FEV1) by 20% following administration of differing concentrations of albuterol (or placebo) by inhalation.

CONTACTS AND LOCATIONS:
Overall Officials: Pai-Chien Chou, MD, PhD, Principal Investigator — Taipei Medical University Hospital
Locations (12):
- India (8):
  - Dr. Jivraj Mehta Smarak Health Foundation, Ahmedabad
  - KLEs Dr Prabhakar Kore Hospital & MRC, Belagāve
  - NRS Medical College and Hospital, Kolkata
  - Medical College and Hospital, Kolkata
  - Aakash Healthcare Super Specialty Hospital, New Delhi
  - Pimpri Chinchwad Municipal Corporation Post Graduate Institute Yashwantrao Chavan Memorial Hospital, Pune
  - Kothrud Hospital, Pune
  - Ashirwad Hospital and Research Centre, Ulhasnagar
- Taiwan (4):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Tamshui Mackay Memorial Hospital, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei